CLINICAL TRIAL: NCT04052841
Title: Automated Morphological Analysis of Meibomian Glands
Brief Title: Morphological Analysis of Meibomian Glands
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Principal Investigator, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190722
Record Dates: First submitted 2019-07-30; First posted 2019-08-12 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: The recruitment of subjects must meet the diagnosis criteria of MGD the international workshop on meibomian gland dysfunction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- MGD-thermal pulsation group (Experimental): A 12 minutes LIPIFLOW treatment was performed.
  Interventions: Procedure: Thermal pulsation
- MGD-IPL group (Experimental): IPL was performed every 3 weeks，3 times in total (0, 3w, 6w).
  Interventions: Procedure: Intense pulsed light therapy
- MGD-manual warm compresses (Experimental): Manual warm compresses were performed every 2 weeks，5 times in total (0, 2w, 4w, 6w, 8w).
  Interventions: Procedure: Manual warm compresses
- Normal health subject group (No Intervention): Normal health subject without intervention.

INTERVENTIONS:
Procedure: Thermal pulsation — Participants underwent a single LipiFlow® thermal pulsation system (TearScience Inc., Morrisville, NC,USA) treatment on the first visit: after lid hygiene with wet cotton swabs(OCuSOFT, Inc., Texas, USA) and instillation of anesthetic eye drops (Alcaine, proparacaine hydrochloride 0.4 ml/2mg) in both eyes, sterile eye cups were placed on to the conjunctival sac as instructed by the manufacturer, after 12 minutes of upper and lower palpebral conjunctival surfaces heat while simultaneously graded pulsatile pressure applying, eye cups were removed slightly.
  Arms: MGD-thermal pulsation group
Procedure: Intense pulsed light therapy — Lid hygiene with wet cotton swabs(OCuSOFT, Inc., Texas, USA) before treatment. Intense pulsed light (IPL) with a range of wavelength (570 or 620 nm) was performed every 3 weeks，3 times in total (0, 3w, 6w). 10 pulses were transmited from one tragus through nose to the other tragus was a single pass, each treatment needed to do 2 passes. Manual lid massage was done after per IPL treatment.
  Arms: MGD-IPL group
Procedure: Manual warm compresses — Lids hygiene of both eyes with wet cotton swabs(OCuSOFT, Inc., Texas, USA).Commercial heated eye patch was use for 10 min. Manual lid massage every 2 weeks, 5 times in total(0，2w, 4w, 4w, 8w).
  Arms: MGD-manual warm compresses

SUMMARY:
An automated quantitative meibomian gland analyzer based on all kinds of infrared meibomian gland images was develop to obtain more detail in meibomian gland, including width, length, area, signal intensity correlated to the quality of meibum, deformation index and ratio of area of each visible specific gland. The purpose of this study is present as separate sections the following points: (1) to compared the detailed characteristics of meibomian glands in normal subjects, Meibomian gland dysfunction (MGD) patients by the automated quantitative analyzer; (2) to identify the inter-examiner and intra-examiner repeatability of the new technique; (3) to explore the correlation among morphological and functional parameters of meibomian gland and risk factors，clinical symptoms and signs; (4) to explore the sensitivity and specificity of meibomian gland morphological and functional parameters in MGD diagnosis. (5) using morphological and functional parameters as new assessment of MGD severity and efficacy indicators for treatment.

DETAILED DESCRIPTION:
Meibomian glands are essential for maintaining ocular surface health and integrity secrete various lipid components to forms a lipid layer to prevent excessive tear evaporation. Functional disorders of the meibomian glands, referred to today as meibomian gland dysfunction (MGD), are increasingly recognized as a high incidence disease commonly characterized by terminal duct obstruction and/or abnormal glandular secretion, often results in ocular surface epithelium damage, chronic blepharitis and dry eye disease that significantly reduces quality of life. A wide variation of the prevalence of MGD were reported from 0.39% to 69.3%, which is likely due to lack of diagnostic methods. To identify which clinical features are likely to be predictive of progressive disease in MGD may indicate the early diagnosis and proper treatment strategies.

Histologic section through the normal meibomian glands and the obstructed human meibomian gland revealed that obstruction of orifice in MGD could lead to dilation of the central duct, damage of the secretory meibocytes and finally result in atrophy of dilated meibomian glands and glands drop-out. It was thus be accepted that detailed changes of meibomian glands morphology are key signs to diagnose and evaluate the severity of MGD. The detailed changes including dilation, distortion, shortening and loss of visualisation of glands which can be directly observed and visual assessment by the developed of non-contact meibomian gland infrared imaging technology. Quantitative evaluations of meibomian glands were obtain by developing imaging processing techniques. The most common use is the image editing software Image J (National Institute of Health; http://imagej.nih.gov/ij) which can identify the gland region on the image manually by the users and may lead to inter-observer variability. Koh et al., first applied original algorithms to automatically analysed gland loss in meibography images with a manually pre-processing. Reiko et al., then develop an objective and automatic system to measure the meibomian gland area. However, the existing methods of meibomian gland analysis have been limited to clinical use where large number of images needs to be analyzed efficiently due to the inter-observer variability or time-consuming process.

Meanwhile, the existing quantitative morphological parameters obtain by those imaging processing techniques, including percentage of MG drop-out and gland atrophy area, were suggested to not only be advanced stages or terminal changes in MGD, but also occurs as an age-related atrophic process. The early findings of MGD induced by the primary pathologic obstruction including degenerative gland dilation, irregularly shapes of gland and change of meibum quality are still difficult to be evaluated automatically and quantitively from the image. Moreover, the meibomian gland drop-out is still an approximate assessment without specific pattern. Whether the atrophy or loss occur in upper or lower eyelids, central, distal or proximal, total loss of gland or partial loss of gland has the greatest effect on the pathology progress of MGD will be important to identify. Thus, a comprehensive analysis technique to automatically detect multi-information of meibomian gland morphology will benefit the future early diagnosis and management of MGD.

Recently, an automated quantitative meibomian gland analyzer based on all kinds of infrared meibomian gland images was develop to obtain more detail in meibomian gland, including width, length, area, signal intensity correlated to the quality of meibum, deformation index and ratio of area of each visible specific gland. The purpose of this study is present as separate sections the following points: (1) to compared the detailed characteristics of meibomian glands in normal subjects and MGD patients by the automated quantitative analyzer; (2) to identify the inter-examiner and intra-examiner repeatability of the new technique; (3) to explore the correlation among morphological and functional parameters of meibomian gland and risk factors，clinical symptoms and signs; (4) to explore the sensitivity and specificity of meibomian gland morphological and functional parameters in MGD diagnosis. (5) using morphological and functional parameters as new assessment of MGD severity and efficacy indicators for treatment.

ELIGIBILITY:
General Inclusion Criteria:

* Age from 18 to 70 years.
* Patients and healthy volunteers who are willing and capable to participate in this clinical study with signed Informed Consent Form.

Inclusion Criteria of patients:

* Clinical diagnosis of MGD: The diagnosis of MGD was based on an altered quality of expressed secretions and/or decreased or absent expression.
* Patients without ≥2/3 Meibomian glands atrophy.
* Fitzpatrick skin type 1-4.

Inclusion Criteria of healthy volunteers:

* Negative history or condition of ocular or systemic illness based on evaluation by a research physician.

General Exclusion Criteria:

* Patients and healthy volunteers with ocular allergies, trauma, contact lens wear, continuous medications usage such as tretinoin, isotretinoin, antidepressant medications, photosensitive drugs, glucocorticoids and immunomodulators, or have used them within one month.
* Patients and healthy volunteers who have a history of ocular surface surgery.
* Patients and healthy volunteers who have active ocular surface infection or have suffered from ocular surface infection within one month.
* Patients and healthy volunteers who have endophthalmitis or a medical history of endophthalmitis.
* Patients and healthy volunteers who have a medical history of viral keratitis infection.
* Women who are pregnant, planning to become pregnant during the course of the study or breast-feeding (women of child-bearing age will be asked by the physician).
* Meibography images were blurred or with obvious tarsus folds, incomplete exposure and large hyperreflective area.
* Patients and healthy volunteers who are not suitable for the trial as determined by investigators.

Exclusion Criteria of patients:

* Patients have abnormalities of ocular surface function or eyelid function, or presence of precancerous lesions, cancer or pigmentation in the eyelid area.
* Patients who have plans to receive ocular surgeries (e.g., cataract, myopic refractive surgery) within 6 months.
* Patients who have been treated with lacrimal punctum embolization within one month.
* Patients with disease that could lead to ADDE, such as Sjogren syndrome and a lacrimal gland abnormality.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Mophology of meibomian glands | 30 days after commencement of treatment
  Infrared photography of inversed upper meibomian glands were measured by Meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany). The infrared images of Meibography were analysed using the new developed software for identifying the mophology features of meibomian glands in millimeter.
Functional feature of meibomian glands | 30 days after commencement of treatment
  Infrared photography of inversed upper and lower meibomian glands were measured by Meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany). The infrared images of Meibography were analysed using the new developed software for identifying the mean signal intensity of meibomian glands in millimeter.

SECONDARY OUTCOMES:
Non-invasive tear-film break-up time | Baseline
  Non-invasived tear-film break-up time is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) with a scale of seconds. Higher values represent a better outcome
Non-invasive tear-film break-up time | 15 days after commencement of treatment
  Non-invasived tear-film break-up time is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) with a scale of seconds. Higher values represent a better outcome
Non-invasive tear-film break-up time | 30 days after commencement of treatment
  Non-invasived tear-film break-up time is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) with a scale of seconds. Higher values represent a better outcome
Non-invasive tear-film break-up time | 90 days after commencement of treatment
  Non-invasived tear-film break-up time is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) with a scale of seconds. Higher values represent a better outcome
Non-invasive tear-film break-up time | 180 days after commencement of treatment
  Non-invasived tear-film break-up time is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) with a scale of seconds. Higher values represent a better outcome
Non-invasive tear meniscus height | Baseline
  Non-invasived tear meniscus height is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) in millimeter. The value higher than 0.20 mm was provided as a normal condition of tear secretion.
Non-invasive tear meniscus height | 15 days after commencement of treatment
  Non-invasived tear meniscus height is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) in millimeter. The value higher than 0.20 mm was provided as a normal condition of tear secretion.
Non-invasive tear meniscus height | 30 days after commencement of treatment
  Non-invasived tear meniscus height is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) in millimeter. The value higher than 0.20 mm was provided as a normal condition of tear secretion.
Non-invasive tear meniscus height | 90 days after commencement of treatment
  Non-invasived tear meniscus height is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) in millimeter. The value higher than 0.20 mm was provided as a normal condition of tear secretion.
Non-invasive tear meniscus height | 180 days after commencement of treatment
  Non-invasived tear meniscus height is measured by tear film pattern of Keratograph 5M (Oculus, Wetzlar, Germany) in millimeter. The value higher than 0.20 mm was provided as a normal condition of tear secretion.
Tear film lipid layer thicknesses | Baseline
  Tear film lipid layer thicknesses were averaged in nanometer(0-100nm) during 20 seconds by LipiView II (Tear Science, Morrisville, NC).
Tear film lipid layer thicknesses | 15 days after commencement of treatment
  Tear film lipid layer thicknesses were averaged in nanometer(0-100nm) during 20 seconds by LipiView II (Tear Science, Morrisville, NC).
Tear film lipid layer thicknesses | 30 days after commencement of treatment
  Tear film lipid layer thicknesses were averaged in nanometer(0-100nm) during 20 seconds by LipiView II (Tear Science, Morrisville, NC).
Tear film lipid layer thicknesses | 90 days after commencement of treatment
  Tear film lipid layer thicknesses were averaged in nanometer(0-100nm) during 20 seconds by LipiView II (Tear Science, Morrisville, NC).
Tear film lipid layer thicknesses | 180 days after commencement of treatment
  Tear film lipid layer thicknesses were averaged in nanometer(0-100nm) during 20 seconds by LipiView II (Tear Science, Morrisville, NC).
The pattern of eye blinks | Baseline
  The pattern of eye blinks including numbers of incompleted and completed blinks during 20 seconds were measured by LipiView II (Tear Science, Morrisville, NC).
The pattern of eye blinks | 15 days after commencement of treatment
  Tear film lipid layer thicknesses and numbers of incomplete blinks during 20 seconds were measured by LipiView II (Tear Science, Morrisville, NC).
The pattern of eye blinks | 30 days after commencement of treatment
  Tear film lipid layer thicknesses and numbers of incomplete blinks during 20 seconds were measured by LipiView II (Tear Science, Morrisville, NC).
The pattern of eye blinks | 90 days after commencement of treatment
  Tear film lipid layer thicknesses and numbers of incomplete blinks during 20 seconds were measured by LipiView II (Tear Science, Morrisville, NC).
The pattern of eye blinks | 180 days after commencement of treatment
  Tear film lipid layer thicknesses and numbers of incomplete blinks during 20 seconds were measured by LipiView II (Tear Science, Morrisville, NC).
Lid margin signs | baseline
  Three lid margin abnormalities (irregular lid margin, plugging of meibomian gland orifices, and anterior or posterior replacement of the mucocutaneous junction) were scored from 0 through 4 according to the number of these abnormalities that were present in each eye. Higher scores represent a worse outcome.
Lid margin signs | 15 days after commencement of treatment
  Three lid margin abnormalities (irregular lid margin, plugging of meibomian gland orifices, and anterior or posterior replacement of the mucocutaneous junction) were scored from 0 through 4 according to the number of these abnormalities that were present in each eye. Higher scores represent a worse outcome.
Lid margin signs | 30 days after commencement of treatment
  Three lid margin abnormalities (irregular lid margin, plugging of meibomian gland orifices, and anterior or posterior replacement of the mucocutaneous junction) were scored from 0 through 4 according to the number of these abnormalities that were present in each eye. Higher scores represent a worse outcome.
Lid margin signs | 90 days after commencement of treatment
  Three lid margin abnormalities (irregular lid margin, plugging of meibomian gland orifices, and anterior or posterior replacement of the mucocutaneous junction) were scored from 0 through 4 according to the number of these abnormalities that were present in each eye. Higher scores represent a worse outcome.
Lid margin signs | 180 days after commencement of treatment
  Three lid margin abnormalities (irregular lid margin, plugging of meibomian gland orifices, and anterior or posterior replacement of the mucocutaneous junction) were scored from 0 through 4 according to the number of these abnormalities that were present in each eye. Higher scores represent a worse outcome.
Meibum expressibility | baseline
  Meibum expressibility were measured by firm digital pressure of Meibomian gland diagnostic Expressibility (Tear Sience, Morrisville, NC):
  For each of these glands, the secretion was graded as follows: 0:no secretion; 1: inspissated/ toothpaste consistency; 2: cloudy liquid secretion and 3: clear liquid secretion19. The scores were then summed in 15 glands to a single meibomian gland yield secretion score (MGYSS) with a range from 0 to 45. Higher values represent a better outcome.
Meibum expressibility | 15 days after commencement of treatment
  Meibum expressibility were measured by firm digital pressure of Meibomian gland diagnostic Expressibility (Tear Sience, Morrisville, NC):
  For each of these glands, the secretion was graded as follows: 0:no secretion; 1: inspissated/ toothpaste consistency; 2: cloudy liquid secretion and 3: clear liquid secretion19. The scores were then summed in 15 glands to a single meibomian gland yield secretion score (MGYSS) with a range from 0 to 45. Higher values represent a better outcome.
Meibum expressibility | 30 days after commencement of treatment
  Meibum expressibility were measured by firm digital pressure of Meibomian gland diagnostic Expressibility (Tear Sience, Morrisville, NC):
  For each of these glands, the secretion was graded as follows: 0:no secretion; 1: inspissated/ toothpaste consistency; 2: cloudy liquid secretion and 3: clear liquid secretion19. The scores were then summed in 15 glands to a single meibomian gland yield secretion score (MGYSS) with a range from 0 to 45. Higher values represent a better outcome.
Meibum expressibility | 90 days after commencement of treatment
  Meibum expressibility were measured by firm digital pressure of Meibomian gland diagnostic Expressibility (Tear Sience, Morrisville, NC):
  For each of these glands, the secretion was graded as follows: 0:no secretion; 1: inspissated/ toothpaste consistency; 2: cloudy liquid secretion and 3: clear liquid secretion19. The scores were then summed in 15 glands to a single meibomian gland yield secretion score (MGYSS) with a range from 0 to 45. Higher values represent a better outcome.
Meibum expressibility | 180 days after commencement of treatment
  Meibum expressibility were measured by firm digital pressure of Meibomian gland diagnostic Expressibility (Tear Sience, Morrisville, NC):
  For each of these glands, the secretion was graded as follows: 0:no secretion; 1: inspissated/ toothpaste consistency; 2: cloudy liquid secretion and 3: clear liquid secretion19. The scores were then summed in 15 glands to a single meibomian gland yield secretion score (MGYSS) with a range from 0 to 45. Higher values represent a better outcome.
Corneal Fluorescein Staining | baseline
  Fluorescein was administered into the conjunctival sac under a cobalt blue light from the slit lamp. Corneal epithelial cell disruption was measured via corneal staining (National Eye Institute (NEI) scale (0-3 scale for each area of 5 areas, total score 15). Higher values represent a worse outcome.
Corneal Fluorescein Staining | 15 days after commencement of treatment
  Fluorescein was administered into the conjunctival sac under a cobalt blue light from the slit lamp. Corneal epithelial cell disruption was measured via corneal staining (National Eye Institute (NEI) scale (0-3 scale for each area of 5 areas, total score 15). Higher values represent a worse outcome.
Corneal Fluorescein Staining | 30 days after commencement of treatment
  Fluorescein was administered into the conjunctival sac under a cobalt blue light from the slit lamp. Corneal epithelial cell disruption was measured via corneal staining (National Eye Institute (NEI) scale (0-3 scale for each area of 5 areas, total score 15). Higher values represent a worse outcome.
Corneal Fluorescein Staining | 90 days after commencement of treatment
  Fluorescein was administered into the conjunctival sac under a cobalt blue light from the slit lamp. Corneal epithelial cell disruption was measured via corneal staining (National Eye Institute (NEI) scale (0-3 scale for each area of 5 areas, total score 15). Higher values represent a worse outcome.
Corneal Fluorescein Staining | 180 days after commencement of treatment
  Fluorescein was administered into the conjunctival sac under a cobalt blue light from the slit lamp. Corneal epithelial cell disruption was measured via corneal staining (National Eye Institute (NEI) scale (0-3 scale for each area of 5 areas, total score 15). Higher values represent a worse outcome.
Schirmer I test | baseline
  The tear production was measured with Schirmer strips without anaesthesia 15 minutes after corneal staining.
Schirmer I test | 15 days after commencement of treatment
  The tear production was measured with Schirmer strips without anaesthesia 15 minutes after corneal staining.
Schirmer I test | 30 days after commencement of treatment
  The tear production was measured with Schirmer strips without anaesthesia 15 minutes after corneal staining.
Schirmer I test | 90 days after commencement of treatment
  The tear production was measured with Schirmer strips without anaesthesia 15 minutes after corneal staining.
Schirmer I test | 180 days after commencement of treatment
  The tear production was measured with Schirmer strips without anaesthesia 15 minutes after corneal staining.
Mophology of meibomian glands | 15 days after commencement of treatment
  Infrared photography of inversed upper meibomian glands were measured by Meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany). The infrared images of Meibography were analysed using the new developed software for identifying the mophology features of meibomian glands in millimeter.
Mophology of meibomian glands | 90 days after commencement of treatment
  Infrared photography of inversed upper meibomian glands were measured by Meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany). The infrared images of Meibography were analysed using the new developed software for identifying the mophology features of meibomian glands in millimeter.
Mophology of meibomian glands | 180 days after commencement of treatment
  Infrared photography of inversed upper meibomian glands were measured by Meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany). The infrared images of Meibography were analysed using the new developed software for identifying the mophology features of meibomian glands in millimeter.
Mophology of meibomian glands | Baseline
  Infrared photography of inversed upper meibomian glands were measured by Meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany). The infrared images of Meibography were analysed using the new developed software for identifying the mophology features of meibomian glands in millimeter.
Functional feature of meibomian glands | Baseline
  Infrared photography of inversed upper and lower meibomian glands were measured by Meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany). The infrared images of Meibography were analysed using the new developed software for identifying the mean signal intensity of meibomian glands in millimeter.
Functional feature of meibomian glands | 15 days after commencement of treatment
  Infrared photography of inversed upper and lower meibomian glands were measured by Meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany). The infrared images of Meibography were analysed using the new developed software for identifying the mean signal intensity of meibomian glands in millimeter.
Functional feature of meibomian glands | 90 days after commencement of treatment
  Infrared photography of inversed upper and lower meibomian glands were measured by Meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany). The infrared images of Meibography were analysed using the new developed software for identifying the mean signal intensity of meibomian glands in millimeter.
Functional feature of meibomian glands | 180 days after commencement of treatment
  Infrared photography of inversed upper and lower meibomian glands were measured by Meibography pattern of Keratograph 5M (Oculus, Wetzlar, Germany). The infrared images of Meibography were analysed using the new developed software for identifying the mean signal intensity of meibomian glands in millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yuan, PHD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (2):
- China (2):
  - Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong
  - Deng Yuqing, Guangzhou

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Supporting Information: Study Protocol

REFERENCES:
- [Result] Arita R, Suehiro J, Haraguchi T, Shirakawa R, Tokoro H, Amano S. Objective image analysis of the meibomian gland area. Br J Ophthalmol. 2014 Jun;98(6):746-55. doi: 10.1136/bjophthalmol-2012-303014. Epub 2013 Jun 27. PMID 23813417
- [Result] Nelson JD, Shimazaki J, Benitez-del-Castillo JM, Craig JP, McCulley JP, Den S, Foulks GN. The international workshop on meibomian gland dysfunction: report of the definition and classification subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1930-7. doi: 10.1167/iovs.10-6997b. Print 2011 Mar. No abstract available. PMID 21450914
- [Result] Schein OD, Munoz B, Tielsch JM, Bandeen-Roche K, West S. Prevalence of dry eye among the elderly. Am J Ophthalmol. 1997 Dec;124(6):723-8. doi: 10.1016/s0002-9394(14)71688-5. PMID 9402817
- [Result] Lekhanont K, Rojanaporn D, Chuck RS, Vongthongsri A. Prevalence of dry eye in Bangkok, Thailand. Cornea. 2006 Dec;25(10):1162-7. doi: 10.1097/01.ico.0000244875.92879.1a. PMID 17172891
- [Result] Uchino M, Dogru M, Yagi Y, Goto E, Tomita M, Kon T, Saiki M, Matsumoto Y, Uchino Y, Yokoi N, Kinoshita S, Tsubota K. The features of dry eye disease in a Japanese elderly population. Optom Vis Sci. 2006 Nov;83(11):797-802. doi: 10.1097/01.opx.0000232814.39651.fa. PMID 17106406
- [Result] Chia EM, Mitchell P, Rochtchina E, Lee AJ, Maroun R, Wang JJ. Prevalence and associations of dry eye syndrome in an older population: the Blue Mountains Eye Study. Clin Exp Ophthalmol. 2003 Jun;31(3):229-32. doi: 10.1046/j.1442-9071.2003.00634.x. PMID 12786773
- [Result] Schaumberg DA, Sullivan DA, Buring JE, Dana MR. Prevalence of dry eye syndrome among US women. Am J Ophthalmol. 2003 Aug;136(2):318-26. doi: 10.1016/s0002-9394(03)00218-6. PMID 12888056
- [Result] Wise RJ, Sobel RK, Allen RC. Meibography: A review of techniques and technologies. Saudi J Ophthalmol. 2012 Oct;26(4):349-56. doi: 10.1016/j.sjopt.2012.08.007. PMID 23961019
- [Result] Tomlinson A, Bron AJ, Korb DR, Amano S, Paugh JR, Pearce EI, Yee R, Yokoi N, Arita R, Dogru M. The international workshop on meibomian gland dysfunction: report of the diagnosis subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2006-49. doi: 10.1167/iovs.10-6997f. Print 2011 Mar. No abstract available. PMID 21450918
- [Result] Simcock B. The role of the intrauterine device in contraceptive practice. Aust Fam Physician. 1976 Mar;5(2):124-39. PMID 942338
- [Result] Knop E, Knop N, Brewitt H, Pleyer U, Rieck P, Seitz B, Schirra F. [Meibomian glands : part III. Dysfunction - argument for a discrete disease entity and as an important cause of dry eye]. Ophthalmologe. 2009 Nov;106(11):966-79. doi: 10.1007/s00347-009-2043-9. German. PMID 19941140
- [Result] Arita R, Itoh K, Maeda S, Maeda K, Furuta A, Fukuoka S, Tomidokoro A, Amano S. Proposed diagnostic criteria for obstructive meibomian gland dysfunction. Ophthalmology. 2009 Nov;116(11):2058-63.e1. doi: 10.1016/j.ophtha.2009.04.037. Epub 2009 Sep 10. PMID 19744718
- [Result] Koh YW, Celik T, Lee HK, Petznick A, Tong L. Detection of meibomian glands and classification of meibography images. J Biomed Opt. 2012 Aug;17(8):086008. doi: 10.1117/1.JBO.17.8.086008. PMID 23224195
- [Result] Knop E, Knop N, Millar T, Obata H, Sullivan DA. The international workshop on meibomian gland dysfunction: report of the subcommittee on anatomy, physiology, and pathophysiology of the meibomian gland. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1938-78. doi: 10.1167/iovs.10-6997c. Print 2011 Mar. No abstract available. PMID 21450915